CLINICAL TRIAL: NCT05603806
Title: Exploring Rheumatoid Arthritis Patients' Disease Activity Using Patient Reported Outcome Measures and Biometric Sensor Data (WEarables Activity in Patients With Rheumatoid Arthritis)
Brief Title: The ArthritisPower Wearable Study
Acronym: WEAR
Status: Completed | Type: Observational
Sponsor: Global Healthy Living Foundation (Other)
Collaborators: University of Alabama at Birmingham (Other); Illumination Health (Network)
Responsible Party: Sponsor
Other Study IDs: Pro00047954
Record Dates: First submitted 2022-09-22; First posted 2022-11-03 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
Keywords: patient-reported outcomes; rheumatoid arthritis; real world evidence; wearable digital technology; real world data; rheumatology; patients; patient-generated health data; mobile technology
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- RA new treatment starts: Adult rheumatoid arthritis patients starting treatment on adalimumab or upadacitinib

SUMMARY:
Rheumatoid arthritis patients being seen at one of the participating clinical sites in a U.S. network of community rheumatology practices who are starting treatment on adalimumab or upadacitinib will be enrolled into a 24-week study combining clinical data from physicians, self-reported patient outcomes from the ArthritisPower registry app, and activity and sleep data from a Fitbit wearable device.

The primary objective of this study is:

• Evaluate longitudinal associations between biometric sensor data (activity and sleep measures), physician-derived data (including clinical disease activity index (CDAI), Rheumatoid Factor (RF) lab results and other relevant biomarkers, current medications and disease duration), and patient-reported outcomes (PROs) (including PROMIS pain interference, physical function, fatigue, sleep disturbance, satisfaction with participation in discretionary social activities, and anxiety).

The secondary objectives of this study are as follows:

* Explore the reliability and predictive validity of biometric sensor data to classify changes in RA disease activity and associated symptoms, including PROs.
* To assess adherence and predictors of adherence with use of biometric sensor
* Assess/track changes in upadacitinib and adalimumab patients using combined physician, PRO and biosensor data.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and above who are adults (i.e., the age of majority where they reside)
* Diagnosis of RA by a physician (as indicated by survey screening questions)
* Currently being seen by a U.S. rheumatologist
* Starting on the day of enrollment (with no prior use ever) or soon-to-initiate (i.e. in the next 28 days) upadacitinib or adalimumab for RA
* Ability to walk without the use of assistive devices;
* Have access to a computer or smartphone to take health assessments and a survey;
* Already own a smartphone (iPhone or Android); iPhone 4S and later or Android 4.3 and later
* Are willing to join the ArthritisPower patient registry;
* Are willing to download the ArthritisPower app;
* Are willing to contribute daily and weekly ePROs for at least at 89 days, and health activity tracker data for at least 84 days (lead-in period minimum of 5 days plus main study period 84 days). Some participants may contribute data more than 89 days if there was a lag in receiving their medication and hence later medication start date;
* Are willing to wear the smartwatch while sleeping;
* Are willing to complete the 7-day run-in requirements (i.e. completing daily PRO assessments for at least 5 of 7 days);
* Have started their medication within 30 days of enrolling in the study (i.e. enrolling in ArthritisPower)
* Will not be out of internet access (wifi and/or mobile data) for 4 or more consecutive days during the study; and
* Willing to be contacted by e-mail/text message and/or phone by the study coordinator if participants fail to adhere to the study Protocol or for any study related assistance as required.
* Clinician must collect a CDAI (including the raw scores for the four components - patient global, physician global and tender and swollen joint count) on day of enrollment.
* CDAI must be >10
* Must have rheumatoid and CCP antibody lab results available, or collect those labs (as part of standard of care during the enrollment visit) if not available

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit patients from non-academic clinical settings and the American Arthritis and Rheumatology Associates (AARA) physician network, Bendcare. All patients seen and treated by Bendcare AARA clinicians may participate in this study should they fit the eligibility criteria. Physicians at these sites will identify patients for their coordinators to enroll. All participants must be or must become ArthritisPower members in order to be eligible for this study consistent with Investigator previously approved studies.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Correlations between patient reported outcomes (PROs), wearable data, and physician derived data | PROs and Wearable Data is collected daily. Physician Derived outcomes are collected at baseline and at follow up appointment at 2-6 months post baseline.
  Pearson correlation coefficient between patient reported outcomes, wearable data, and physician derived data PROs include:Daily- Pain NRS 0-10; Fatigue NRS 0-10; Duration of Morning Joint Stiffness Weekly- Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5); Patient Global Assessment; PROMIS Pain Interference CAT; PROMIS Physical Function CAT; PROMIS Fatigue CAT; PROMIS Sleep Disturbance CAT Monthly- PROMIS Satisfaction with Participation in Discretionary Social Activities; PROMIS Anxiety Wearable Data include:Activity- steps, distance, energy expenditure, metabolic equivalents, time walking per day, time in activity intensity per day, active time, aerobic time Heart rate-beats per minute, time in heart rate zones; Sleep-time asleep/restless/awake, and derived variables.
  Physician derived outcomes include:Clinical Disease Activity Index (CDAI); RA Clinical Labs (Rheumatoid Factor lab results); Current prescription medications for RA; Years since RA diagnosis

SECONDARY OUTCOMES:
Changes in RA disease activity and associated symptoms | CDAI is collected at baseline and then again at a follow up appointment from 2-6 months after baseline.
  Changes in RA will be measured using change in Clinical Disease Activity Index (CDAI) between baseline and follow up visits
Adherence to PRO measures | PROs Data is collected daily for up to 6 months
  Adherence*: percent of days completing ePROs
Adherence to wearing Fitbit | Wearable Data is collected daily for up to 6 months
  Adherence*: percent of days wearing Fitbit
Predictors of adherence | PROs and Wearable Data is collected daily for up to 6 months
  Using Patient Reported Outcomes and wearable data to predict who is adherent to study protocol
  PROs include:Daily- Pain NRS 0-10; Fatigue NRS 0-10; Duration of Morning Joint Stiffness Weekly- Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5); Patient Global Assessment; PROMIS Pain Interference CAT; PROMIS Physical Function CAT; PROMIS Fatigue CAT; PROMIS Sleep Disturbance CAT Monthly- PROMIS Satisfaction with Participation in Discretionary Social Activities; PROMIS Anxiety Wearable Data include:Activity- steps, distance, energy expenditure, metabolic equivalents, time walking per day, time in activity intensity per day, active time, aerobic time Heart rate-beats per minute, time in heart rate zones; Sleep-time asleep/restless/awake, and derived variables.
Changes in upadacitinib and adalimumab patients using combined physician, PRO and biosensor data. | PROs Data is collected daily from baseline physician appointment until follow up appointment. Physician derived outcomes are collected at baseline and then again at a follow up appointment from 2-6 months after baseline.
  Changes will be measured using numerical scales for PROs.
  PROs include:Daily- Pain NRS 0-10; Fatigue NRS 0-10; Duration of Morning Joint Stiffness Weekly- Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5); Patient Global Assessment; PROMIS Pain Interference CAT; PROMIS Physical Function CAT; PROMIS Fatigue CAT; PROMIS Sleep Disturbance CAT Monthly- PROMIS Satisfaction with Participation in Discretionary Social Activities; PROMIS Anxiety Wearable Data include:Activity- steps, distance, energy expenditure, metabolic equivalents, time walking per day, time in activity intensity per day, active time, aerobic time Heart rate-beats per minute, time in heart rate zones; Sleep-time asleep/restless/awake, and derived variables.
  Physician derived outcomes include:Clinical Disease Activity Index (CDAI); RA Clinical Labs (Rheumatoid Factor lab results); Current prescription medications for RA; Years since RA diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Laura Stradford, MPH, Principal Investigator — Global Healthy Living Foundation
Locations (1):
- Global Healthy Living Foundation, Upper Nyack, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowell WB, Curtis JR, Nolot SK, Curtis D, Venkatachalam S, Owensby JK, Poon JL, Calvin AB, Kannowski CL, Faries DE, Gavigan K, Haynes VS. Digital Tracking of Rheumatoid Arthritis Longitudinally (DIGITAL) Using Biosensor and Patient-Reported Outcome Data: Protocol for a Real-World Study. JMIR Res Protoc. 2019 Sep 26;8(9):e14665. doi: 10.2196/14665. PMID 31573949
- [Background] Nowell WB, Curtis D, Thai M, Wiedmeyer C, Gavigan K, Venkatachalam S, Ginsberg S, Curtis JR. Digital Interventions to Build a Patient Registry for Rheumatology Research. Rheum Dis Clin North Am. 2019 May;45(2):173-186. doi: 10.1016/j.rdc.2019.01.009. PMID 30952391
- [Background] Nowell WB, Curtis JR, Crow-Hercher R. Patient Governance in a Patient-Powered Research Network for Adult Rheumatologic Conditions. Med Care. 2018 Oct;56 Suppl 10 Suppl 1(10 Suppl 1):S16-S21. doi: 10.1097/MLR.0000000000000814. PMID 30074946
- [Background] Yun H, Nowell WB, Curtis D, H Willig J, Yang S, Auriemma M, Chen L, Filby C, Curtis JR. Assessing Rheumatoid Arthritis Disease Activity With Patient-Reported Outcomes Measurement Information System Measures Using Digital Technology. Arthritis Care Res (Hoboken). 2020 Apr;72(4):553-560. doi: 10.1002/acr.23888. PMID 30927515
- See also: ArthritisPower — http://arthritispower.org